CLINICAL TRIAL: NCT04023097
Title: Self-selection Study to Confirm the "Toothwave" Labeling and User Manual Are Clear Enough for Contraindicated Users to Self-exclude Themselves From Using the Device
Brief Title: Self-selection Study of the Toothwave Toothbrush
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Home Skinovations Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: DO116508
Record Dates: First submitted 2019-07-11; First posted 2019-07-17 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2019-07

CONDITIONS: Gingivitis; Plaque; Calculus; Tooth Discoloration
MeSH Terms: conditions — Gingivitis; Plaque, Amyloid; Calculi; Tooth Discoloration

STUDY DESIGN:
Intervention Model Description: 5 participants are suppose to exclude themselves from the use of the device, while the 5 others should claim they can use it.
Who Masked: Participant
Masking Description: Before they start their part in the study, participants won't be aware if they can use the brush or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Toothwave contraindicated subject (Experimental): the Toothwave toothbrush is contraindicated for people in certain conditions, e.g. pregnant or nursing women, people with pacemaker and more.
  This arm is assembled from contraindicated subject, who should exclude themselves from use of the device, based on the user manual and box sleeve.
  Interventions: Device: Toothwave toothbrush
- potential users of the Toothwave device (Active Comparator): The control arm is assembled from people who can use the toothbrush and should recognize themselves as potential users.
  Interventions: Device: Toothwave toothbrush

INTERVENTIONS:
Device: Toothwave toothbrush — Subjects get the device's box with the user manual and the device. However, they don't use the device, but only read the user manual and fill questionnaires.

SUMMARY:
This study objective is to test the Silk'n Toothwave self-selection, by potential end users. Additionally, this study will evaluate if contraindicated subjects will self-exclude from use of the device and the ability to understand accurately the labeling content (box and user manual).

DETAILED DESCRIPTION:
The Silk'n Toothwave Device, in its original packaging, along with the user manual will be provided to the patient in a simulated home use environment. The patient labeling will be in the format intended for distribution.

All subjects will sign an informed consent before any study activity. Five (5) potential end users and Additional five (5) contraindicated subjects will be screened for this self-selection study. Subjects will be provided with the device in its original packaging and will be evaluated for their ability to decide if they are eligible or they should self-exclude themselves from use of the device based solely on reading the device labeling (box and user manual).

Once the subjects complete reviewing the labeling materials (box and user manual) they will be requested to perform a labeling comprehension exam for testing the ability to correctly understand the labeling content.

The study will not include treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female equal to or greater than 18 years of age.
2. Subject is a potential candidate for purchasing the Silk'n Toothwave Device.
3. Subject is capable of understanding and is willing to sign informed consent.

Exclusion Criteria:

1. Current or history of oral cavity cancer or oropharyngeal cancer.
2. Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body.
3. Pregnant or nursing.
4. Any active condition in the oral cavity at the discretion of the investigator.
5. Any surgery in the oral cavity within 3 months prior to treatment, or before complete healing.

Modified Inclusion Criteria for contraindicated subjects:

1. Subject with or an active implant, such as a pacemaker, incontinence device, insulin pump, etc.
2. Subject is pregnant or nursing (lactating).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Subjects will mention in the post-reading questionnaire if they should use the Toothwave device or not. | 30 minutes
  Post-reading questionnaire includes the question: "are you allowed to use this device?". Based on reading the user manual and box labeling, subjects should answer "yes" or "no" according to their condition.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Hellman, MD, Principal Investigator — Hellman Dermatology Clinic
Locations (1):
- Hellman Dermatology clinic, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No